CLINICAL TRIAL: NCT04006847
Title: Effect of Omega-3 Fatty Acid, Eicosapentaenoic Acid, and Its Metabolites in Combination With Tyrosine Kinase Inhibitors in Chronic Myeloid Leukemia in Stable Chronic Phase
Brief Title: Omega -3 Fatty Acid in Combination With Tyrosine Kinase Inhibitors in Chronic Myeloid Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Product complaint
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Seema Naik, MD, Assistant Professor, Cancer Institutue, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 17-085
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Results first posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Chronic Myeloid Leukemia, Chronic Phase
Keywords: Omega-3 Fatty Acid; Eicosapentaenoic Acid; Tyrosine Kinase Inhibitors; TKI; GoldAID Eicosapentaenoic Acid; Fish Oil
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — Eicosapentaenoic Acid; Fatty Acids, Omega-3; Tyrosine Kinase Inhibitors; Imatinib Mesylate; Dasatinib; nilotinib; bosutinib

STUDY DESIGN:
Intervention Model Description: Phase I/II, open-label, single site study using a standard 3 + 3 statistical design to determine the MTD and the recommended Phase 2 dose for oral EPA when administered to subjects receiving on a TKI pre-study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Eicosapentaenoic Acid (EPA) (Experimental): Phase I: TKI with escalating/de-escalating doses of EPA to determine MTD.
  Phase I dose levels: Dose Level 1 = EPA 1500 mg orally once per day; Dose Level 2 = EPA 2000 mg orally once per day; Dose Level 3 = EPA 3000 mg orally once per day; Dose Level -1 = EPA 1000 mg orally once per day; Dose Level -2 = EPA 500 mg orally once per day.
  Phase II: TKI administered in combination with the recommended Phase II dose of EPA
  Interventions: Drug: Eicosapentaenoic Acid; Drug: Tyrosine kinase inhibitor

INTERVENTIONS:
Drug: Eicosapentaenoic Acid — Eicosapentaenoic Acid once per day orally
  Other Names: Omega-3 fatty acid
Drug: Tyrosine kinase inhibitor — Tyrosine kinase inhibitor to be administered at subjects' pre-study dose
  Other Names: TKI; Imatinib; Dasatinib; Nilotinib; Bosutinib

SUMMARY:
This is a Phase I/II single site, open label clinical trial. The purpose of the Phase I portion is to determine the safety, tolerability, and recommended Phase II dose of Eicosapentaenoic Acid (EPA) when given daily in combination with a Tyrosine Kinase Inhibitor (TKI) in subjects with Chronic Myeloid Leukemia (CML) in chronic stable phase. The recommended Phase II dose will be the maximum tolerated dose (MTD) of EPA as determined by the evaluation of dose-limiting toxicities (DLTs). The Phase II portion will subsequently examine the Anti-CML effects of EPA when administered with a TKI at the recommended Phase II dose. This efficacy objective will be done by evaluating BCR-ABL p210 quantitative PCR blood levels every 3 months to 1 year.

DETAILED DESCRIPTION:
Targeting CML leukemia stem cells is of paramount importance in successfully preventing cancer relapse. EPA metabolite, Δ12-PGJ3 may represent a new chemotherapeutic agent for leukemia that targets leukemia stem cells. Selective targeting of cancer stem cells may be potentially a highly effective treatment for cancer. As most CML patients treated with a TKI will reach a complete cytogenetic response, quantification of residual BCR-ABL transcripts by quantitative reverse transcription PCR (RT-qPCR) is a critical tool to further monitor response kinetics. Addition of EPA to TKI may help decrease residual BCR-ABL positive (Ph+) leukemia stem cells.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age.
2. Confirmed diagnosis of CML ≥ 18 months from diagnosis.
3. Current concomitant treatment with TKI therapy (Imatinib, Dasatinib, Nilotinib or Bosutinib; excluding Ponatinib). TKI therapy should be stable (same drug and dose) for at least 3 months prior to study enrollment.
4. One of the following confirmed:

   1. BCR-ABL p210 at stable molecular disease (e.g., MMR stable but not CMR)
   2. HR but no MMR.
5. Stable molecular response defined as 2 sequential BCR-ABL p210 levels done in the same lab with less than ½ log reduction of BCR-ABL (BA) 3-6 months apart.
6. ECOG PS of ≤ 3
7. Adequate organ function, as defined by the following:

   ANC ≥ 500 cells/mm3 Platelet count ≥ 50,000 cells/mm3 Serum bilirubin ≤ 1.5 x ULN AST and ALT ≤ 2.5 x ULN Alkaline phosphatase ≤ 2.5 x ULN
8. WOCP as defined as defined as not surgically sterile or not one year post-menopausal, must have a negative result for a serum or urine pregnancy test within 7 days of initial receipt of study drug. Surgically sterile is defined as having had a hysterectomy, tubal ligation, or oophorectomy.
9. WOCP must use a medically accepted method of contraception and must agree to continued use of this method for the duration of the study and for 30 days after last dose of study drug. Acceptable methods of contraception include abstinence, barrier method with spermicide, intrauterine device (IUD) known to have a failure rate of less than 1% per year, or steroidal contraceptive (oral, transdermal, implanted, or injected) in conjunction with a barrier method.
10. Male subjects capable of producing offspring, must use a medically accepted method of birth control and agree to continued use of this method for the duration of the study and for 30 days after last dose of study drug because of the possible effects on spermatogenesis. Acceptable methods of contraception include abstinence, barrier method with spermicide, WOCP partner's use of an IUD known to have a failure rate of less than 1% per year, WOCP partner's use of steroidal contraceptive (oral, implanted or injected) in conjunction with a barrier method, WOCP partner is surgically sterile or 1 year postmenopausal. In addition, male subjects may not donate sperm for the duration of the study and for 30 days after last dose of study drug.

Exclusion Criteria:

1. Has a malignancy or infection requiring active treatment
2. Has a known HIV infection, Hepatitis B , or Hepatitis C infection
3. Has a known symptomatic congestive heart failure (CHF), unstable angina or cardiac arrhythmia
4. Is using Aspirin or NSAID or COX-I
5. Is known to be non-compliant to medications.
6. Has, in the opinion of the physician investigator, an uncontrolled medical or psychiatric disorder.
7. Has active central nervous system (CNS) leukemia.
8. Is preceding allogeneic stem HSCT.
9. Has a known T 315 I mutation.
10. Is taking FISH oil at EPA dose > 500 mg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seema Naik, MD, Principal Investigator — Penn State Cancer Institute
Locations (1):
- Penn State Cancer Institute, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject was consented but withdrew from participation.
Groups:
- Eicosapentaenoic Acid (EPA): Phase I: TKI with escalating/de-escalating doses of EPA to determine MTD.
  Phase I dose levels: Dose Level 1 = EPA 1500 mg orally once per day; Dose Level 2 = EPA 2000 mg orally once per day; Dose Level 3 = EPA 3000 mg orally once per day; Dose Level -1 = EPA 1000 mg orally once per day; Dose Level -2 = EPA 500 mg orally once per day.
  Phase II: TKI administered in combination with the recommended Phase II dose of EPA
  Eicosapentaenoic Acid: Eicosapentaenoic Acid once per day orally
  Tyrosine kinase inhibitor: Tyrosine kinase inhibitor to be administered at subjects' pre-study dose
Period: Overall Study
Arm/Group | Eicosapentaenoic Acid (EPA)
Started | 1
Completed | 0
Not Completed | 1
Not completed — Product issue | 1

BASELINE CHARACTERISTICS:
Arm/Group | Eicosapentaenoic Acid (EPA)
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase I - Recommended Phase II Dose of EPA
Description: Recommended Phase II dose of EPA will be established by using a standard 3 + 3 statistical design to determine the MTD as assessed by DLTs when administered orally in combination with a TKI in subjects with CML in stable chronic phase. Toxicity will be evaluated using the NCI Common Toxicity Criteria (CTC) version 5.0.
Time Frame: the time of initiation of the study medication to 30 days after last dose of study medication
Population: data were not collected
Groups:
- Eicosapentaenoic Acid (EPA): Phase I: TKI with escalating/de-escalating doses of EPA to determine MTD.
  Phase I dose level: Dose Level 1 = EPA 1500 mg orally once per day;
Arm/Group | Eicosapentaenoic Acid (EPA)
Number analyzed (Participants) | 0

2. Primary Outcome: Phase II - Anti-CML Response to Recommended Phase II Dose Eicosapentaenoic Acid
Description: BCR-ABL transcript levels will be assessed every 3 months post initiation of Eicosapentaenoic Acid to assess Anti-CML response.
Time Frame: 1 year
Population: data were not collected
Arm/Group | Eicosapentaenoic Acid (EPA)
Number analyzed (Participants) | 0

3. Secondary Outcome: Molecular Responses of CML
Description: Log reduction from stable molecular response with bcr-abl PCR at MR 3 or more to bcr-abl to major molecular response (MR 4.5) or complete molecular response
Time Frame: 1 year
Population: data were not collected
Arm/Group | Eicosapentaenoic Acid (EPA)
Number analyzed (Participants) | 0

4. Secondary Outcome: Induction of Apoptosis in CML Leukemia Stem Cell by Formation of Δ12-PGJ3 and Other Metabolites
Description: Apoptosis will be analyzed by in vitro correlative studies using subject's plasma with effect on known leukemia cell line with CML leukemic stem cells. EPA metabolite will be examined by flow cytometry using Annexin V staining and adding serum from treated study subject to murine CML cells grown in vitro culture. The evaluation will be done at baseline, Month 1, and every 3 months up to year 2
Time Frame: 2 years
Population: data were not collected
Arm/Group | Eicosapentaenoic Acid (EPA)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: CTCAE v. 5.0
Arm/Group | Eicosapentaenoic Acid (EPA)
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Due to the product issues, the trials was halted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-19): https://cdn.clinicaltrials.gov/large-docs/47/NCT04006847/Prot_SAP_000.pdf